CLINICAL TRIAL: NCT00943098
Title: Efficacy and Safety of a Single s.c. Diclofenac HPBCD 75mg/1ml Injection as Compared to a Single i.m. Voltarol® 75mg/3ml, in the Treatment of Acute Moderate-to-severe Post-surgical Pain Following Dental Surgery (Impacted 3rd Molar Removal).
Brief Title: Evaluation of the Efficacy and Safety of Diclofenac HPBCD 75mg/ml in Treatment of Pain Following Dental Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IBSA Institut Biochimique SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09PUK-DCsc05
Record Dates: First submitted 2009-07-21; First posted 2009-07-22 (Estimated); Results first posted 2013-01-28 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2012-12

CONDITIONS: Dental Pain
MeSH Terms: conditions — Toothache | interventions — Diclofenac

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diclofenac HPBCD s.c. 75mg/ml (Experimental)
  Interventions: Drug: Diclofenac HPBCD s.c. 75mg/ml
- Voltarol 75mg/3ml i.m. (Active Comparator)
  Interventions: Drug: Voltarol 75mg/3ml i.m.

INTERVENTIONS:
Drug: Diclofenac HPBCD s.c. 75mg/ml — 1 single injection at day of dental surgical extraction
  Arms: Diclofenac HPBCD s.c. 75mg/ml
Drug: Voltarol 75mg/3ml i.m. — 1 single injection at day of dental surgical extraction
  Arms: Voltarol 75mg/3ml i.m.

SUMMARY:
The present study is aimed at demonstrating the therapeutic equivalence of diclofenac HPBCD 75mg/1ml s.c. with the marketed reference product, Voltarol® 75mg/3ml i.m. in the treatment of acute moderate-to-severe pain after dental impaction surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgical extraction of a single fully or partially impacted mandibular 3rd molar requiring bone removal.
* Patients experiencing moderate to severe post-operative pain within 6 hours from end of surgery.
* Pre-operative laboratory tests in the reference ranges or without clinically significant abnormalities as judged by the Investigator.

Exclusion Criteria:

* Surgery performed under general anaesthesia, or sedation.
* Complications occurring during the surgical procedure or in the period before randomisation as judged by the investigator.
* Acute local or systemic infection at the time of surgery that could confound the post-surgical evaluation.
* Patients with clinical signs of gastritis, gastro-duodenal ulcer, GI bleeding. Other GI disturbances or disease that in the opinion of the investigator could be negatively affected by the administration of NSAIDs.
* Clinical signs or history of coagulation disorders that could be negatively affected by NSAIDs administration.
* Hepatic or renal impairment.
* Patients with significant cardiac impairment, history of cerebrovascular disease, history or peripheral arterial disease, uncontrolled hypertension.
* Hypersensitivity to diclofenac or other NSAIDs or to one of the study medication components.
* Patients under chronic treatment with topical or systemic analgesics/NSAIDs.
* Patients under treatment with any medication that may affect the treatment efficacy evaluation.
* Patients under treatment with any medication whose concomitant use may be susceptible to interactions with diclofenac or may affect safety.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2009-09; Primary Completion 2010-03 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian Brook, Prof, Principal Investigator — The school of Clinical Dentistry
Locations (3):
- United Kingdom (3):
  - The School of Dentistry, University of Birmingham, Birmingham
  - Department of oral Surgery; University Dental Hospital, Cardiff
  - The School of Clinical Dentistry, The University of Sheffield, Sheffield

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients already scheduled for the surgical extraction of a single fully or partially impacted mandibular 3rd molar requiring bone removal underwent a screening visit within 30 days from the scheduled date of surgery.
Groups:
- Diclofenac HPBCD s.c. 75mg/ml: Diclofenac HPBCD s.c. 75mg/ml : 1 single injection at day of dental surgical extraction
- Voltarol 75mg/3ml i.m.: Voltarol 75mg/3ml i.m. : 1 single injection at day of dental surgical extraction
Period: Overall Study
Arm/Group | Diclofenac HPBCD s.c. 75mg/ml | Voltarol 75mg/3ml i.m.
Started | 70 | 72 (1 patient was excluded from the ITT and therefore the baseline population is 71)
Completed | 70 | 72
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diclofenac HPBCD s.c. 75mg/ml | Voltarol 75mg/3ml i.m. | Total
Number analyzed (Participants) | 70 | 71 | 141
Age Continuous [Mean (Standard Deviation); unit: years] | 28.1 (6.88) | 28.7 (7.08) | 28.49 (6.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 32 | 74
  Male | 28 | 39 | 67

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity Difference (PID)
Description: Pain intensity difference (PID) was derived by subtracting each pain intensity score (PI) from the baseline PI score (t0), where PI was assessed by the patient on a 0-100 mm VAS (from 0 = no pain to 100 = worst pain imaginable).
Time Frame: 1.5 hours
Population: Analysed patients are those included in the PP population: all patients included in the ITT population who also met all inclusion/exclusion criteria and who did not have any major protocol violation, and with post-surgical pain assessment at the primary endpoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: mm
Arm/Group | Diclofenac HPBCD s.c. 75mg/ml | Voltarol 75mg/3ml i.m.
Number analyzed (Participants) | 64 | 65
mm | 44.8 (40.5 to 49.1) [40.5 to 49.1] | 45.5 [41.2 to 49.8]
Statistical Analysis 1: Comparison: Diclofenac HPBCD s.c. 75mg/ml vs Voltarol 75mg/3ml i.m; Assuming a difference in means of 0 mm, a common standard deviation of 22.5 mm, a sample size of 60 subjects in each group had 95% power to reject the null hypothesis; Test type: Non-Inferiority or Equivalence — The sample size calculation was based on a hypothesis of non-inferiority of Diclofenac HPBCD 75mg/ml s.c. versus Voltarol® 75mg/3ml i.m. with regard to the primary efficacy variable (PID at 1.5 hours after study drug administration). The clinically significant difference (delta) between groups was defined in 15 mm of pain intensity difference (a 30% decline from starting levels of pain intensity of 50 mm or greater on a 0 to 100 VAS); p = 0.813, ANCOVA; Mean Difference (Final Values) = -0.71, 95% CI 2-sided [-6.62 to 5.20]

2. Secondary Outcome: PIDs
Time Frame: at 15 minutes post-dose.
Population: Analysed patients were included in the ITT population: all randomized patients who received the study medication and with at least one post-baseline efficacy evaluation within 1.5 hours post-dose (primary endpoint).
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Diclofenac HPBCD s.c. 75mg/ml | Voltarol 75mg/3ml i.m.
Number analyzed (Participants) | 70 | 71
mm | 7.37 (13.1) | 6.83 (15.6)

3. Secondary Outcome: PIDs
Time Frame: at 30 minutes post-dose.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Diclofenac HPBCD s.c. 75mg/ml | Voltarol 75mg/3ml i.m.
Number analyzed (Participants) | 70 | 71
mm | 19.8 (17.1) | 18.4 (18.9)

4. Secondary Outcome: PIDs
Time Frame: at 45 minutes post-dose.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Diclofenac HPBCD s.c. 75mg/ml | Voltarol 75mg/3ml i.m.
Number analyzed (Participants) | 70 | 71
mm | 31.2 (18.8) | 37.9 (19.6)

5. Secondary Outcome: PIDs
Time Frame: at 60 minutes post-dose.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Diclofenac HPBCD s.c. 75mg/ml | Voltarol 75mg/3ml i.m.
Number analyzed (Participants) | 70 | 71
mm | 37.6 (18.8) | 37.9 (19.6)

6. Secondary Outcome: PIDs
Time Frame: at 90 minutes post-dose.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Diclofenac HPBCD s.c. 75mg/ml | Voltarol 75mg/3ml i.m.
Number analyzed (Participants) | 70 | 71
mm | 44.0 (18.4) | 45.0 (17.9)

7. Secondary Outcome: PIDs
Time Frame: at 2 hours post-dose.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Diclofenac HPBCD s.c. 75mg/ml | Voltarol 75mg/3ml i.m.
Number analyzed (Participants) | 70 | 71
mm | 49.0 (16.0) | 50.3 (16.1)

8. Secondary Outcome: PIDs
Time Frame: at 3 hours post-dose.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Diclofenac HPBCD s.c. 75mg/ml | Voltarol 75mg/3ml i.m.
Number analyzed (Participants) | 70 | 71
mm | 49.7 (17.0) | 53.3 (15.0)

9. Secondary Outcome: PIDs
Time Frame: at 4 hours post-dose.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Diclofenac HPBCD s.c. 75mg/ml | Voltarol 75mg/3ml i.m.
Number analyzed (Participants) | 70 | 71
mm | 50.6 (14.6) | 53.9 (15.5)

10. Secondary Outcome: PIDs
Time Frame: at 5 hours post-dose.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Diclofenac HPBCD s.c. 75mg/ml | Voltarol 75mg/3ml i.m.
Number analyzed (Participants) | 70 | 71
mm | 48.7 (15.7) | 52.3 (15.6)

11. Secondary Outcome: PIDs
Time Frame: at 6 hours post-dose.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Diclofenac HPBCD s.c. 75mg/ml | Voltarol 75mg/3ml i.m.
Number analyzed (Participants) | 70 | 71
mm | 47.5 (14.4) | 51.2 (16.3)

12. Secondary Outcome: PIDs
Time Frame: at 7 hours post-dose.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Diclofenac HPBCD s.c. 75mg/ml | Voltarol 75mg/3ml i.m.
Number analyzed (Participants) | 70 | 71
mm | 42.8 (17.2) | 49.6 (18.2)

13. Secondary Outcome: PIDs
Time Frame: at 8 hours post-dose.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Diclofenac HPBCD s.c. 75mg/ml | Voltarol 75mg/3ml i.m.
Number analyzed (Participants) | 70 | 71
mm | 43.7 (15.8) | 47.1 (17.9)

14. Primary Outcome: Pain Intensity Difference (PID)
Description: as for outcome 1
Time Frame: 1.5 hours
Population: Analysed patients are those included in the ITT population: defined as all randomised patients who received the study medication and with at least one post-baseline efficacy evaluation within 1.5 hours post-dose.
Measure: Least Squares Mean (95% Confidence Interval); unit: mm
Arm/Group | Diclofenac HPBCD s.c. 75mg/ml | Voltarol 75mg/3ml i.m.
Number analyzed (Participants) | 70 | 71
mm | 44.2 [40.0 to 48.3] | 44.7 [40.6 to 48.8]
Statistical Analysis 1: Comparison: Diclofenac HPBCD s.c. 75mg/ml vs Voltarol 75mg/3ml i.m; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.862, ANCOVA; Mean Difference (Final Values) = -0.51, 95% CI 2-sided [-6.23 to 5.22]

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the signature o fthe informed consent to study end.
Arm/Group | Diclofenac HPBCD s.c. 75mg/ml | Voltarol 75mg/3ml i.m.
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/72
Other Adverse Events (participants affected / at risk) | 49/70 | 41/72
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diclofenac HPBCD s.c. 75mg/ml (N=70) | Voltarol 75mg/3ml i.m. (N=72)
Nausea (Gastrointestinal disorders) | 13 (14) | 3 (3)
Vomiting (Gastrointestinal disorders) | 5 (5) | 0 (0)
injection site haematoma (General disorders) | 12 (12) | 4 (4)
Injection site pain (General disorders) | 11 (11) | 8 (8)
Injection site reaction (General disorders) | 7 (7) | 8 (8)
Alveolar osteitis (Infections and infestations) | 6 (7) | 4 (4)
Nasopharyngitis (Infections and infestations) | 2 (2) | 4 (4)
wound infection (Infections and infestations) | 3 (3) | 5 (5)
Headache (Nervous system disorders) | 11 (12) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less